CLINICAL TRIAL: NCT02872870
Title: Developmental Language Difficulties: Behavioural and Electrophysiological Studies of the Connections Between Spoken and Written Language and Specificity of These Disorders
Brief Title: Developmental Language Difficulties: Behavioural and Electrophysiological Studies
Acronym: LANGAGE
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: Université de Lille 3 (Unknown); Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0020
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Dyslexia; Dysphasia
Keywords: language disorders; developmental disorders of oral and written language
MeSH Terms: conditions — Dyslexia; Aphasia; Language Disorders | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control adults: lexical tests and electroencephalogram (EEG).
  Interventions: Behavioral: auditory lexical decision task; Device: electroencephalogram
- Dyslexic patients: lexical tests
  Interventions: Behavioral: auditory lexical decision task; Device: electroencephalogram
- Dysphasic patients: lexical tests
  Interventions: Behavioral: auditory lexical decision task; Device: electroencephalogram

INTERVENTIONS:
Behavioral: auditory lexical decision task
Device: electroencephalogram

SUMMARY:
This study will help to better characterize oral and written language disorders and determine if these disorders are continuous or not. The participants ( dyslexic and dysphasic patients and control adults) will carry out an auditory lexical decision task during which an electroencephalogram (EEG) will be recorded.

ELIGIBILITY:
Inclusion Criteria (patients):

* Non-verbal intelligence quotient (IQ) less than 85 according to the Wechsler Intelligence Scale for Children (WISC) perceptual index
* Specific oral language disorders diagnosed by the multidisciplinary team (neurologist, psychologist, speech therapist): understanding language deficit, estimated by the test SCOTLAND (Lecocq, 1996) and / or vocabulary test (Dunn Thiébaud).
* Specific written language disorders (dyslexia) diagnosed by a multidisciplinary team according to a test that can objectify the late reading (Alouette) and locate deficits (EVALEC)
* Be affiliated to a social security regimen
* Have signed an informed consent or signed by the parents if the patient is minor
* Aged at least 8 years old

Inclusion Criteria (controls)

* Non-deficit (>85) non-verbal Wechsler Scale (codes and matrices)
* No specific oral language disorders
* No specific written language disorders (dyslexia)
* Be affiliated to a social security regimen
* Have signed an informed consent or signed by the parents if the patient is minor
* Aged at least 8 years old

Exclusion Criteria:

* Mother tongue other than French
* Non-verbal reasoning abilities below 85 measured by the WISC 4 (for patients only) and Non-verbal capacities of reasoning lower than the normal measured by the non-verbal scale of Wechsler (for controls only)
* Presence of pervasive developmental disorders
* No affiliation to a social security regimen
* Absence of signature of the informed consent
* Subject of less than 8 years

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of 3 groups. A group of volunteers (controls), a group of patients with oral language disorders, a group of patients with written language disorders.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Score Alouette reading test | at inclusion
  In this test, the participant has to read in a loud voice a text, during three minutes. The final score takes into account the speed and the number of errors. For test performance, clinical groups will be compared with its controls.
Score EVALEC reading test | at inclusion
  For test performance, clinical groups will be compared with its controls.
Score silence reading test | at inclusion
  A group of letters will be presented and the participant has to say if this letters compose a known word. For test performance, clinical groups will be compared with its controls.
Score of reading comprehension test | at inclusion
  For test performance, clinical groups will be compared with its controls.
Score of Khomsi | at inclusion
  The objective of this group of different tests is to evaluate comprehension and production of oral language. For test performance, clinical groups will be compared with its controls.

SECONDARY OUTCOMES:
Measure of the electroencephalography power spectra | at inclusion
  For test performance, clinical groups will be compared with its controls.
Correlation between electroencephalography power spectra and clinical outcome | at inclusion
  For test performance, clinical groups will be compared with its controls.

CONTACTS AND LOCATIONS:
Overall Officials: Séverine Casalis, Study Director — Université de Lille 3; Françoise Boidein, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille (GHICL)
Locations (3):
- Université catholique de Louvain (IPSY), Louvain-la-Neuve, Belgium
- France (2):
  - Hôpital Saint Vincent de Paul (GHICL), Lille
  - Université de Lille 3 Charles de Gaulle (URECA), Villeneuve-d'Ascq

IPD SHARING:
Plan to Share IPD: No